CLINICAL TRIAL: NCT05396924
Title: Is Rectal Temperature Measurement Quicker in Detecting Hypothermia During Hip Arthroscopy
Brief Title: Rectal Temperature Measurement in Detecting Hypothermia During Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Enejd Veizi, MD, Assistant Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E2-21-862
Record Dates: First submitted 2022-04-06; First posted 2022-05-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Hip Arthropathy; Hypothermia; Orthopedic Disorder
Keywords: femoroacetabular impingement; hip arthroscopy; hypothermia; rectal temperature
MeSH Terms: conditions — Hypothermia; Musculoskeletal Diseases; Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled study with sequential randomization; the first patient will be included in the 1st group, and the second patient will be included into the 2nd group. All patients scheduled for hip arthroscopy during the defined study period are eligible for inclusion. While room temperature irrigation fluids will be used routinely for Group 1, irrigation fluids heated up to 36-38 degrees will be used for the other group. Patients will be operated in the same operating room and at the same room temperature. A probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a thermometer. Mean body temperatures measured from 2 different locations between the groups will be compared, and the probability of detecting early local and later general hypothermia from the rectal mucosa will be examined.
Who Masked: Participant, Investigator
Masking Description: Enrolled patients and investigator of final output data will be blinded to the study protocol. Care providers (surgeons, nurses and OR personnel) will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room Group (Active Comparator): Room temperature irrigation fluids will be used routinely for Group 1. Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer, whose batteries will be changed every two operations.
  Interventions: Procedure: Rectal temperature measurement; Procedure: Temporal temperature measurement
- Warmed Group (Active Comparator): Irrigation fluids heated up to 36-38 degrees will be used for Group 2.Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer, whose batteries will be changed every two operations.
  Interventions: Procedure: Rectal temperature measurement; Procedure: Temporal temperature measurement

INTERVENTIONS:
Procedure: Rectal temperature measurement — Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer. The data obtained will be analyzed by a blinded researcher. Mean body temperatures measured from 2 different locations (temporal region and rectal mucosa) between the groups will be compared, and the probability of detecting early local and later general hypothermia from the rectal mucosa will be examined
Procedure: Temporal temperature measurement — Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer. The data obtained will be analyzed by a blinded researcher. Mean body temperatures measured from 2 different locations (temporal region and rectal mucosa) between the groups will be compared, and the probability of detecting early local and later general hypothermia from the rectal mucosa will be examined

SUMMARY:
Irrigation fluids used during hip arthroscopy surgery are generally stored at room temperature and are cooler than the core temperature of the patient. They are used abundantly during hip arthroscopy surgery. The aim of this study is to detect local and then general hypothermia that may occur by monitoring the body temperature from the rectal mucosa of patients undergoing hip arthroscopy, using irrigation fluids of different temperatures and comparing it with the temperature measured from the temporal region.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study where sequential randomization will be applied to patients; The first patient will be included in the 1st group, and the second patient will be included into the 2nd group, and so on. All patients scheduled for hip arthroscopy in our institution during the defined study period are eligible for inclusion. While room temperature irrigation fluids will be used routinely for Group 1, irrigation fluids heated up to 36-38 degrees will be used for the other group. Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer, whose batteries will be changed every two operations. The data obtained will be analyzed by a blinded researcher. Mean body temperatures measured from 2 different locations (temporal region and rectal mucosa) between the groups will be compared, and the probability of detecting early local and later general hypothermia from the rectal mucosa will be examined.

ELIGIBILITY:
Inclusion Criteria:

- Patients between the ages of 18-50 undergoing hip arthroscopy and willing to participate

Exclusion Criteria:

* Patients with a previous history of surgery from the same hip
* Patients with a history of thyroid disease (hypo/hyperthyroidism)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Is rectal temperature measurement more effective in detecting hypothermia? | During the intervention, every 15 minutes.
  Throughout the intervention, every 15 minutes, temperature will be measured from the rectum and from the temporal region. Rectal temperature measurements will be compared to temporal measurements in a standardized environment (OR room temperature, noted every 15 min). Comparison will show whether rectal temperature measurement is superior to temporal measurement in detecting intraoperative hypothermia during hip arthroscopy.

SECONDARY OUTCOMES:
Does the usage of warmed irrigation fluids avoid or delay intraoperative hypothermia during hip arthroscopy? | During the intervention, every 15 minutes.
  While room temperature irrigation fluids will be used routinely for Group 1, irrigation fluids heated up to 36-38 degrees will be used for the other group. Patients will be operated in the same operating room and at the same room temperature with the same type/amount of covering and body warming. At the start of the surgical procedure, a probe inserted into the rectal mucosa will measure the patient's body temperature every 15 minutes. In addition, the temperature of the patients will be measured from their temporal regions with a contactless thermometer. The secondary outcome of this study is to investigate whether usage of warmed irrigation fluids avoid or delay intraoperative hypothermia during hip arthroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Kasım Kılıçarslan, MD, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital - Ankara Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available at the end of the study for a period of 6 months.

REFERENCES:
- [Background] Parodi D, Valderrama J, Tobar C, Besomi J, Lopez J, Lara J, Ilic JP. Effect of warmed irrigation solution on core body temperature during hip arthroscopy for femoroacetabular impingement. Arthroscopy. 2014 Jan;30(1):36-41. doi: 10.1016/j.arthro.2013.08.035. Epub 2013 Oct 30. PMID 24183196
- [Background] Ukrani RD, Arif A, Sadruddin A, Hasan O, Noordin S. Intraoperative hypothermia in patients undergoing Total knee arthroplasty: a cross-sectional study from a developing country. BMC Musculoskelet Disord. 2021 May 31;22(1):504. doi: 10.1186/s12891-021-04390-7. PMID 34059046
- [Background] Nordgren M, Hernborg O, Hamberg A, Sandstrom E, Larsson G, Soderstrom L. The Effectiveness of Four Intervention Methods for Preventing Inadvertent Perioperative Hypothermia During Total Knee or Total Hip Arthroplasty. AORN J. 2020 Mar;111(3):303-312. doi: 10.1002/aorn.12961. PMID 32128778
- [Background] Ohki K, Kawano R, Yoshida M, Kanosue I, Yamamoto K. Normothermia is Best Achieved by Warming Above and Below with Pre-warming Adjunct: A Comparison of Conductive Fabric Versus Forced-air and Water. Surg Technol Int. 2019 May 15;34:40-45. PMID 31037721
- [Background] Williams M, El-Houdiri Y. Inadvertent hypothermia in hip and knee total joint arthroplasty. J Orthop. 2018 Jan 20;15(1):151-158. doi: 10.1016/j.jor.2018.01.035. eCollection 2018 Mar. PMID 29379254
- [Background] Simpson JB, Thomas VS, Ismaily SK, Muradov PI, Noble PC, Incavo SJ. Hypothermia in Total Joint Arthroplasty: A Wake-Up Call. J Arthroplasty. 2018 Apr;33(4):1012-1018. doi: 10.1016/j.arth.2017.10.057. Epub 2017 Nov 8. PMID 29195854
- [Background] Aksu C, Kus A, Gurkan Y, Solak M, Toker K. Survey on Postoperative Hypothermia Incidence In Operating Theatres of Kocaeli University. Turk J Anaesthesiol Reanim. 2014 Apr;42(2):66-70. doi: 10.5152/TJAR.2014.15010. Epub 2014 Jan 6. PMID 27366393
- [Derived] Firat A, Veizi E, Kalayci I, Sezgin BS, Erdogan Y, Gursoy S, Capurro-Soler B, Koutserimpas C. Heated Irrigation Fluids Did Not Reduce the Prevalence of Rectally Measured Hypothermia During Hip Arthroscopic Surgery Compared With Room-Temperature Fluids: A Prospective Randomized Trial. Orthop J Sports Med. 2025 Jun 26;13(6):23259671251350401. doi: 10.1177/23259671251350401. eCollection 2025 Jun. PMID 40584085